CLINICAL TRIAL: NCT04365270
Title: The Antimicrobial Activity and Clinical Performance of Chitosan-modified Glass Ionomer: A Randomized Clinical Trial
Brief Title: Antibacterial Effect and Clinical Performance of Chitosan Modified Glass Ionomer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar Assem Hodhod, Principal Investigator,Teaching Assistant ,Dentist, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-REC IM 011730
Record Dates: First submitted 2019-12-06; First posted 2020-04-28 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Reversible Pulpitis; Pulpitis; Caries,Dental; Caries Class I; Caries; Dentin; Caries
Keywords: Glass ionomer; Chitosan; Titanium dioxide; Titanium dioxide nanoparticles; Chlorhexidine; indirect pulp capping; Alternative restorative technique; stepwise caries excavation; antibacterial restorative; incomplete caries removal; primary molars; early childhood caries
MeSH Terms: conditions — Pulpitis; Dental Caries | interventions — glass ionomer; fuji IX; Chlorhexidine; titanium dioxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All participants and assessors will be masked,the wil just deal with the randomized numbers.
  except the care provider because the materials consistency before mixing is obvious in 2 of the 3 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chitosan Glass ionomer (Experimental): purified low molecular weight and viscosity chitosan will be dissolved in 0.1 mol/L acetic acid to be used to modify the stock liquid provided with the glassionomer Fuji IX to have 10% v/v chitosan.
  will be placed in the prepared cavity over the last layer of caries
  Interventions: Drug: Glass Ionomer; Drug: Chitosan Low Molecular Weight (20-200 Mpa.S)
- Chitosan/Titanium dioxide nanoparticles Glass ionomer (Experimental): The stock liquid provided with the glassionomer Fuji IX will be modified with 10%v/v purified low molecular weight and viscosity chitosan will be dissolved in 0.1 mol/L acetic acid.
  The Powder will be modified with 3% titanium dioxide nanoparticles will be placed in the prepared cavity over the last layer of caries
  Interventions: Drug: Glass Ionomer; Drug: Chitosan Low Molecular Weight (20-200 Mpa.S); Drug: Titanium Dioxide
- Chlorhexidine glass ionomer (Active Comparator): Chlorhexidine Diacetate will be added to the powder of Fuji IX with 0.5% v/v
  Interventions: Drug: Glass Ionomer; Drug: Chlorhexidine Diacetate
- Glass ionomer (Placebo Comparator): Stock powder and liquid Fuji IX from GC japan
  Interventions: Drug: Glass Ionomer

INTERVENTIONS:
Drug: Glass Ionomer — Glass ionomer filling material would be modified accordingly or used as is
  Other Names: Fuji IX
Drug: Chitosan Low Molecular Weight (20-200 Mpa.S) — deacetylated chitin, poly(D-glucosamine) purified by dissolving in 0.1 mol/L acetic acid, then precipitated in 0.1 mol/L sodium hydroxide and the precipitate will be washed with ethanol/water (70/30 v/v) mixture followed by freeze drying
  Other Names: Aldrich, cat#448869, lot #STBG9041
  Arms: Chitosan Glass ionomer; Chitosan/Titanium dioxide nanoparticles Glass ionomer
Drug: Chlorhexidine Diacetate — Chlorhexidine antibacterial effect to be compared by Sigma-aldrich PHR 1222 , lot#LRAB3716
  Other Names: chlorhexidine acetate
  Arms: Chlorhexidine glass ionomer
Drug: Titanium Dioxide — Titanium(IV) oxide,nanopowder, 21 nm primary particle size (TEM), >99.5% trace metals basis cat#718467 Lot#MKCB6332 Lot #MKCB6332
  Other Names: Titanium(IV) oxide
  Arms: Chitosan/Titanium dioxide nanoparticles Glass ionomer

SUMMARY:
The study is a randomized clinical trial that assesses the clinical success and the antibacterial effect on carious dentine of glass ionomer when modified with Chitosan and/or Titanium dioxide nano particles vs the control group of modification with Chlorhexidine as control when used in primary molars

DETAILED DESCRIPTION:
Participants will be recruited from the acquitted to the clinic of pediatric dentistry department , Faculty of Dentistry of Ain Shams University. random allocation of the participants where indirect pulp capping is indicated so that modified Glass ionomer would be used as the filling material.

partial removal of caries is done then caries sample would be taken and sent for a microbiological evaluation and then, cavity dimensions is recoded, finally placement of the modified glass ionomer in the prepared cavity.

In a total period of 9 months the patients will be followed every 3 months for clinical evaluation and in the final visit the filling would be removed and another bacterial sample would be taken for comparison, then a permanent filling is placed.

ELIGIBILITY:
Inclusion Criteria:

The teeth will be primary molars selected from patients presented to the outpatient clinic that are

* Healthy patients.
* Age: 4-8 years.
* Children having at least one primary molar with only occlusal caries having dentine lesions wide enough for the smallest excavator to enter (Ø=0.9 mm).

Exclusion Criteria:

* Teeth with pulp involvement, those suffering from pain, irreversible pulpits or pulp necrosis.
* Children with systemic diseases.
* Patients with history of active para-functional oral habits, xerostomia.
* Patients who will have difficulties in cooperating.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Antibacterial | 9 months
  Dentin samples incubated on 2 culture mediums and total bacterial count by counting colony forming units will be counted. Higher number means Less antibacterial effect
Clinical performance | followup 9 months
  "Modified United States Public Health Service Ryge Criteria" for Direct Clinical Evaluation and rating of Restoration.measuring color match, anatomic contour, marginal integrity, cavosurface marginal discoloration, secondary caries, surface texture, gross fracture.
  each outcome will be graded Alpha(A) for the highest score, Bravo(b) for moderate score, and Charlie(C) for the lowest score.

CONTACTS AND LOCATIONS:
Overall Officials: Mariem Wassel, Assistant professor, Study Chair — Ainshams University; Noha Kabil, Professor, Study Director — Ainshams university; omar A Hodhod, Dentist, Principal Investigator — British University in cairo
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulder R, Anderson-Small C. Ion release of chitosan and nanodiamond modified glass ionomer restorative cements. Clin Cosmet Investig Dent. 2019 Sep 6;11:313-320. doi: 10.2147/CCIDE.S220089. eCollection 2019. PMID 31686917
- [Background] Wassel MO, Khattab MA. Antibacterial activity against Streptococcus mutans and inhibition of bacterial induced enamel demineralization of propolis, miswak, and chitosan nanoparticles based dental varnishes. J Adv Res. 2017 Jul;8(4):387-392. doi: 10.1016/j.jare.2017.05.006. Epub 2017 May 17. PMID 28560054
- [Result] Ibrahim MA, Meera Priyadarshini B, Neo J, Fawzy AS. Characterization of Chitosan/TiO2 Nano-Powder Modified Glass-Ionomer Cement for Restorative Dental Applications. J Esthet Restor Dent. 2017 Apr;29(2):146-156. doi: 10.1111/jerd.12282. Epub 2017 Feb 12. PMID 28190299
- [Result] Ibrahim MA, Neo J, Esguerra RJ, Fawzy AS. Characterization of antibacterial and adhesion properties of chitosan-modified glass ionomer cement. J Biomater Appl. 2015 Oct;30(4):409-19. doi: 10.1177/0885328215589672. Epub 2015 Jun 15. PMID 26079388
- [Result] Kabil NS, Badran AS, Wassel MO. Effect of the addition of chlorhexidine and miswak extract on the clinical performance and antibacterial properties of conventional glass ionomer: an in vivo study. Int J Paediatr Dent. 2017 Sep;27(5):380-387. doi: 10.1111/ipd.12273. Epub 2016 Oct 21. PMID 27766712